CLINICAL TRIAL: NCT00850200
Title: Improving the Therapeutic Ratio by Using Proton Beam Radiation Therapy for Patients With Stage IA-IIIBX (Bulky/Non-bulky) Hodgkin Lymphoma Involving the Mediastinum Following Standard Chemotherapy
Brief Title: Proton Therapy for Hodgkin Lymphoma
Acronym: HL01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0806 - HL01
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma, Proton Radiation
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proton Radiation Plan (Experimental)
  Interventions: Radiation: Proton Radiation Plan
- Conventional Photon Radiation Plan (Active Comparator)
  Interventions: Radiation: Conventional Photon Radiation Plan
- Intensity Modulated Radiation Plan (Active Comparator)
  Interventions: Radiation: Intensity Modulated Radiation Plan

INTERVENTIONS:
Radiation: Proton Radiation Plan — Between 21-39.6 Gy/CGE to the PTV
  Arms: Proton Radiation Plan
Radiation: Conventional Photon Radiation Plan — Between 21-39.6 Gy/CGE to the PTV
  Arms: Conventional Photon Radiation Plan
Radiation: Intensity Modulated Radiation Plan — Between 21-39.6 Gy/CGE to the PTV
  Arms: Intensity Modulated Radiation Plan

SUMMARY:
The purpose of this study is to reduce the risk of radiation related side effects and complications by treating with radiation (protons or photons) that exposes less of normal organs to low dose radiation.

DETAILED DESCRIPTION:
3 treatment plans will be created to deliver between a total of 21-39.6 Gray (Gy)/Centigray Equivalents (CGE) to the planning target volume (PTV).

1. Proton Plan
2. Conventional Plan
3. Intensity Modulated Radiotherapy (IMRT) Plan

The patient will then receive the radiation modality with the lowest percentage of the body receiving 4 Gy (V4Gy/CGE)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed "classic" Hodgkin lymphoma.
* Completed chemotherapy.

Exclusion Criteria:

* Prior radiotherapy.
* Prior or concurrent cancer other than non-melanomatous skin cancer.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2013-05 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford S Hoppe, MD, MPH, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] Bonadonna G, Bonfante V, Viviani S, Di Russo A, Villani F, Valagussa P. ABVD plus subtotal nodal versus involved-field radiotherapy in early-stage Hodgkin's disease: long-term results. J Clin Oncol. 2004 Jul 15;22(14):2835-41. doi: 10.1200/JCO.2004.12.170. Epub 2004 Jun 15. PMID 15199092
- [Background] Horning SJ, Hoppe RT, Breslin S, Bartlett NL, Brown BW, Rosenberg SA. Stanford V and radiotherapy for locally extensive and advanced Hodgkin's disease: mature results of a prospective clinical trial. J Clin Oncol. 2002 Feb 1;20(3):630-7. doi: 10.1200/JCO.2002.20.3.630. PMID 11821442
- [Background] Straus DJ, Portlock CS, Qin J, Myers J, Zelenetz AD, Moskowitz C, Noy A, Goy A, Yahalom J. Results of a prospective randomized clinical trial of doxorubicin, bleomycin, vinblastine, and dacarbazine (ABVD) followed by radiation therapy (RT) versus ABVD alone for stages I, II, and IIIA nonbulky Hodgkin disease. Blood. 2004 Dec 1;104(12):3483-9. doi: 10.1182/blood-2004-04-1311. Epub 2004 Aug 17. PMID 15315964
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Kawashima T, Hudson MM, Meadows AT, Friedman DL, Marina N, Hobbie W, Kadan-Lottick NS, Schwartz CL, Leisenring W, Robison LL; Childhood Cancer Survivor Study. Chronic health conditions in adult survivors of childhood cancer. N Engl J Med. 2006 Oct 12;355(15):1572-82. doi: 10.1056/NEJMsa060185. PMID 17035650
- [Background] Constine LS, Tarbell N, Hudson MM, Schwartz C, Fisher SG, Muhs AG, Basu SK, Kun LE, Ng A, Mauch P, Sandhu A, Culakova E, Lyman G, Mendenhall N. Subsequent malignancies in children treated for Hodgkin's disease: associations with gender and radiation dose. Int J Radiat Oncol Biol Phys. 2008 Sep 1;72(1):24-33. doi: 10.1016/j.ijrobp.2008.04.067. PMID 18722263
- [Background] van Leeuwen FE, Klokman WJ, Stovall M, Dahler EC, van't Veer MB, Noordijk EM, Crommelin MA, Aleman BM, Broeks A, Gospodarowicz M, Travis LB, Russell NS. Roles of radiation dose, chemotherapy, and hormonal factors in breast cancer following Hodgkin's disease. J Natl Cancer Inst. 2003 Jul 2;95(13):971-80. doi: 10.1093/jnci/95.13.971. PMID 12837833
- [Background] Ng AK, Bernardo MV, Weller E, Backstrand K, Silver B, Marcus KC, Tarbell NJ, Stevenson MA, Friedberg JW, Mauch PM. Second malignancy after Hodgkin disease treated with radiation therapy with or without chemotherapy: long-term risks and risk factors. Blood. 2002 Sep 15;100(6):1989-96. doi: 10.1182/blood-2002-02-0634. PMID 12200357
- [Background] Behringer K, Josting A, Schiller P, Eich HT, Bredenfeld H, Diehl V, Engert A; German Hodgkin Lymphoma Study Group. Solid tumors in patients treated for Hodgkin's disease: a report from the German Hodgkin Lymphoma Study Group. Ann Oncol. 2004 Jul;15(7):1079-85. doi: 10.1093/annonc/mdh273. PMID 15205202
- [Background] Campbell BA, Voss N, Pickles T, Morris J, Gascoyne RD, Savage KJ, Connors JM. Involved-nodal radiation therapy as a component of combination therapy for limited-stage Hodgkin's lymphoma: a question of field size. J Clin Oncol. 2008 Nov 10;26(32):5170-4. doi: 10.1200/JCO.2007.15.1001. Epub 2008 Oct 6. PMID 18838714
- [Background] Girinsky T, Pichenot C, Beaudre A, Ghalibafian M, Lefkopoulos D. Is intensity-modulated radiotherapy better than conventional radiation treatment and three-dimensional conformal radiotherapy for mediastinal masses in patients with Hodgkin's disease, and is there a role for beam orientation optimization and dose constraints assigned to virtual volumes? Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):218-26. doi: 10.1016/j.ijrobp.2005.06.004. Epub 2005 Sep 19. PMID 16169675
- [Background] Goodman KA, Toner S, Hunt M, Wu EJ, Yahalom J. Intensity-modulated radiotherapy for lymphoma involving the mediastinum. Int J Radiat Oncol Biol Phys. 2005 May 1;62(1):198-206. doi: 10.1016/j.ijrobp.2004.08.048. PMID 15850922
- [Background] Nieder C, Schill S, Kneschaurek P, Molls M. Influence of different treatment techniques on radiation dose to the LAD coronary artery. Radiat Oncol. 2007 Jun 5;2:20. doi: 10.1186/1748-717X-2-20. PMID 17547777
- [Background] Schneider U, Lomax A, Lombriser N. Comparative risk assessment of secondary cancer incidence after treatment of Hodgkin's disease with photon and proton radiation. Radiat Res. 2000 Oct;154(4):382-8. doi: 10.1667/0033-7587(2000)154[0382:craosc]2.0.co;2. PMID 11023601
- [Background] Sigurdson AJ, Ronckers CM, Mertens AC, Stovall M, Smith SA, Liu Y, Berkow RL, Hammond S, Neglia JP, Meadows AT, Sklar CA, Robison LL, Inskip PD. Primary thyroid cancer after a first tumour in childhood (the Childhood Cancer Survivor Study): a nested case-control study. Lancet. 2005 Jun 11-17;365(9476):2014-23. doi: 10.1016/S0140-6736(05)66695-0. PMID 15950715
- [Background] Nieder C, Schill S, Kneschaurek P, Molls M. Comparison of three different mediastinal radiotherapy techniques in female patients: Impact on heart sparing and dose to the breasts. Radiother Oncol. 2007 Mar;82(3):301-7. doi: 10.1016/j.radonc.2006.10.015. Epub 2006 Dec 6. PMID 17156873
- [Background] Travis LB, Gospodarowicz M, Curtis RE, Clarke EA, Andersson M, Glimelius B, Joensuu T, Lynch CF, van Leeuwen FE, Holowaty E, Storm H, Glimelius I, Pukkala E, Stovall M, Fraumeni JF Jr, Boice JD Jr, Gilbert E. Lung cancer following chemotherapy and radiotherapy for Hodgkin's disease. J Natl Cancer Inst. 2002 Feb 6;94(3):182-92. doi: 10.1093/jnci/94.3.182. PMID 11830608
- [Background] Travis LB, Hill DA, Dores GM, Gospodarowicz M, van Leeuwen FE, Holowaty E, Glimelius B, Andersson M, Wiklund T, Lynch CF, Van't Veer MB, Glimelius I, Storm H, Pukkala E, Stovall M, Curtis R, Boice JD Jr, Gilbert E. Breast cancer following radiotherapy and chemotherapy among young women with Hodgkin disease. JAMA. 2003 Jul 23;290(4):465-75. doi: 10.1001/jama.290.4.465. PMID 12876089
- [Background] Graham MV, Purdy JA, Emami B, Harms W, Bosch W, Lockett MA, Perez CA. Clinical dose-volume histogram analysis for pneumonitis after 3D treatment for non-small cell lung cancer (NSCLC). Int J Radiat Oncol Biol Phys. 1999 Sep 1;45(2):323-9. doi: 10.1016/s0360-3016(99)00183-2. PMID 10487552
- [Background] Tsujino K, Hirota S, Endo M, Obayashi K, Kotani Y, Satouchi M, Kado T, Takada Y. Predictive value of dose-volume histogram parameters for predicting radiation pneumonitis after concurrent chemoradiation for lung cancer. Int J Radiat Oncol Biol Phys. 2003 Jan 1;55(1):110-5. doi: 10.1016/s0360-3016(02)03807-5. PMID 12504042
- [Background] Hernando ML, Marks LB, Bentel GC, Zhou SM, Hollis D, Das SK, Fan M, Munley MT, Shafman TD, Anscher MS, Lind PA. Radiation-induced pulmonary toxicity: a dose-volume histogram analysis in 201 patients with lung cancer. Int J Radiat Oncol Biol Phys. 2001 Nov 1;51(3):650-9. doi: 10.1016/s0360-3016(01)01685-6. PMID 11597805
- [Background] Bhatia S, Robison LL, Oberlin O, Greenberg M, Bunin G, Fossati-Bellani F, Meadows AT. Breast cancer and other second neoplasms after childhood Hodgkin's disease. N Engl J Med. 1996 Mar 21;334(12):745-51. doi: 10.1056/NEJM199603213341201. PMID 8592547
- [Background] Eich HT, Haverkamp U, Engert A, Kocher M, Skripnitchenko R, Brillant C, Sehlen S, Duhmke E, Diehl V, Muller RP. Biophysical analysis of the acute toxicity of radiotherapy in Hodgkin's lymphoma--a comparison between extended field and involved field radiotherapy based on the data of the German Hodgkin Study Group. Int J Radiat Oncol Biol Phys. 2005 Nov 1;63(3):860-5. doi: 10.1016/j.ijrobp.2005.02.053. Epub 2005 May 31. PMID 15925455
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] IRB #70-2003: Radiation Oncology Outcome Tracking Project (RADTRAC); PI: Robert J. Amdur.

RESULTS

PARTICIPANT FLOW:
Groups:
- Optimal Treatment Plan: Each patient has three radiation treatment plans conducted prior to initiation of treatment (proton, IMRT, conventional). Only the plan that's found to be the most optimal in regard to minimizing the heart v4 is the one that was actually used to treat the patient. In this case, the proton plan was found to be the optimal plan in each case; patients were therefore treated with proton therapy between 21-39.6 Gray (Gy)/Centigray Equivalents (CGE) to the planning target volume (PTV).
  The primary endpoint of this study is the paired differences among the three plans. Thus there's just one treatment arm.
Period: Overall Study
Arm/Group | Optimal Treatment Plan
Started | 20
Completed | 15
Not Completed | 5
Not completed — Physician Decision | 2
Not completed — Did not recieve treatment | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 20 patients were enrolled. One decided to withdrawal after being enrolled, but prior to any treatment plans being performed.
Groups:
- Proton Therapy Plan Compared to IMRT and Conventional RT: Each patient has a proton, IMRT and conventional plan done prior to treatment for dosimetric comparison of the primary endpoint which is the percent of the body that receives 4 Gray (%V4). The plan that delivers the smallest %V4 will be the plan that is pursued for actual treatment. Therefore, each patient will have three treatment plans, but will only be treated with one of these three plans (the superior one).
Arm/Group | Proton Therapy Plan Compared to IMRT and Conventional RT
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 24.5 (13.5) [7.7 to 57.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Normal Tissue Exposed to Greater Than or Equal to 4 Gy/CGE With Use of Proton Therapy Compared to Both Intensity Modulated Radiotherapy (IMRT) and Conventional Therapy.
Time Frame: Immediately proceeding completion of each of the three treatment plans
Measure: Median (Full Range); unit: percentage of body receiving 4 Gy
Arm/Group | Proton Radiation Plan | Conventional Photon Radiation Plan | Intensity Modulated Radiation Plan
Number analyzed (Participants) | 19 | 19 | 19
percentage of body receiving 4 Gy | 0.161 [0.062 to 0.346] | 0.291 [0.162 to 0.497] | 0.355 [0.189 to 0.811]

2. Secondary Outcome: Percentage of Participants Who Survived
Description: Overall survival as assessed with the Kaplan-Meier product limit method.
Time Frame: 4 years after beginning of radiation therapy
Population: Patients treated with the optimal dosimetric modality
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Treated Cohort: Overall survival as estimated with the Kaplan-Meier product limit method at 4 years after treatment.
Arm/Group | Treated Cohort
Number analyzed (Participants) | 15
percentage of participants | 92 [61 to 99]

3. Secondary Outcome: Percentage of Participants Who Did Not Have Disease Progression
Description: Disease free survival as assessed with the Kaplan-Meier product limit method
Time Frame: 4 years after beginning of radiation therapy
Population: Patients treated with the optimal dosimetric modality
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treated Cohort
Number analyzed (Participants) | 15
percentage of participants | 93 [63 to 99]

ADVERSE EVENTS:
Time Frame: Cumulative adverse events were collected via regular 6 month patient follow-ups after the completion of treatment.
Description: There were 20 patients initially enrolled. One decided to not receive treatment after initial enrollment. Three had treatment plans completed (and thus contributed that data), but sought treatment elsewhere. One patient was withdrawn after treatment. There are therefore only 15 of 20 enrolled patients actually assessable for adverse events.
Groups:
- Superior Treatment Plan: Each patient has three radiation treatment plans conducted prior to initiation of treatment (proton, IMRT, conventional). Only the plan that's found to be the most optimal in regard to minimizing the heart v4 is the one that was actually used to treat the patient. In this case, the proton plan was found to be the optimal plan in each case; patients were therefore treated with proton therapy between 21-39.6 Gray (Gy)/Centigray Equivalents (CGE) to the planning target volume (PTV).
  The primary endpoint of this study is the paired differences among the three plans. Thus there's just one treatment arm.
Arm/Group | Superior Treatment Plan
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Superior Treatment Plan (N=15)
Dyspepsia - acute grade 2 (Gastrointestinal disorders) | 3 (3)
Esophagitis - acute grade 2 (Gastrointestinal disorders) | 3 (3)
Skin toxicity - grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
thyroid problem - grade 2 (Endocrine disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes